CLINICAL TRIAL: NCT01178034
Title: Early Identification of Warfarin Maintenance Dose in Patients With Atrial Fibrillation: a Randomized Trial Evaluating a New Genotype-based Versus Usual Care Initiation of Treatment
Brief Title: Early Identification of Warfarin Maintenance Dosage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Vittorio Pengo, Professor of Cardiology, University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1643P
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Atrial Fibrillation
Keywords: Warfarin; Dose; Pharmacogenetic; INR
MeSH Terms: conditions — Atrial Fibrillation | interventions — Genetic Algorithms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pharmacogenetic warfarin dose (Experimental): Warfarin maintenance dose on the basis of demographic/pharmacogenetic data
  Interventions: Genetic: Calculate warfarin dose using demographic/genetic algorithm

INTERVENTIONS:
Genetic: Calculate warfarin dose using demographic/genetic algorithm — Age, body weight and genetic to calculate warfarin dosage

SUMMARY:
Initiation of warfarin therapy is problematic. The investigators goal was to evaluate if a new demographic/pharmacogenetic algorithm is better than a usual algorithm based on INR value at day five after four days of 5 mg/day warfarin. To this end patients with atrial fibrillation starting warfarin are randomized in two arms.

DETAILED DESCRIPTION:
The objective of this randomized study is to evaluate the accuracy of a new demographic/pharmacogenetic as compared to usual warfarin dosing algorithm in predicting warfarin maintenance dose. In patients with atrial fibrillation starting anticoagulation, the loading dose of warfarin in the tested group is calculated on the basis of VKORC1 genotype and patient's body weight.The second day warfarin maintenance dose is calculated on the basis of surface area and CYP2C9, CYP4F2 e VKORC1 genotype. In the usual care group the maintenance dose at day 5 is calculated on the basis of a published algorithm (Pengo V, Am J Cardiol 2001). INR is checked on day 0, 5, 7, 9, 12, 15 and 19. Primary end-point of the trial is the number of INR outside the therapeutic range of 2.0 to 3.0. Secondary end-points are the number of changes in dose prescription, the difference between predicted and actual warfarin maintenance dose and thrombotic and bleeding events.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Indication to warfarin with INR between 2.0 and 3.0

Exclusion Criteria:

* Pregnancy
* Drug interactions
* Basal INR > 1.2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
International Normalized Ratio (INR) | Day 0, 5, 7, 9, 12, 15, 19.
  Number of INR outside the therapeutic range (INR 2.0-3.0)

SECONDARY OUTCOMES:
Number of changes in warfarin dosage | Day 0-19
Difference between predicted and actual warfarin maintenance dose | Day 19
Thromboembolic and Bleeding complications | Day 0-30

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Pengo, M.D., Principal Investigator — University of Padova
Locations (1):
- Thrombosis Centre, Padua, Italy

REFERENCES:
- [Derived] Pengo V, Zambon CF, Fogar P, Padoan A, Nante G, Pelloso M, Moz S, Frigo AC, Groppa F, Bozzato D, Tiso E, Gnatta E, Denas G, Padayattil Jose S, Padrini R, Basso D, Plebani M. A Randomized Trial of Pharmacogenetic Warfarin Dosing in Naive Patients with Non-Valvular Atrial Fibrillation. PLoS One. 2015 Dec 28;10(12):e0145318. doi: 10.1371/journal.pone.0145318. eCollection 2015. PMID 26710337